CLINICAL TRIAL: NCT00354939
Title: 10-week, Open, National, Multicenter Clinical Trial to Evaluate the Safety of Insulin Glargine in Type 2 Diabetes Mellitus Patients, on Intensified Conventional Therapy (ICT)
Brief Title: Insulin Analogue With Continuous Glucose Monitoring System (CGMS) Measurement
Acronym: SAFIR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HOE901_4049
Record Dates: First submitted 2006-07-19; First posted 2006-07-20 (Estimated); Last update posted 2010-08-31 (Estimated); Status verified 2010-08

CONDITIONS: Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine

INTERVENTIONS:
Drug: Insulin glargine

SUMMARY:
Primary objective:

Difference in frequency of subjects with conventionally detected hypoglycemia by the subject [at least one measurement smaller/equal 60mg/dl documented in the 8-point profile in the case record form (CRF) or documentation of symptomatic hypoglycemia in the CRF through Visits 8/9] compared to CGMS detected blood glucose values smaller/equal 60mg/dl during CGMS measurements (at least one measurement through Visits 8/9) after eight weeks of treatment with insulin glargine.

Secondary objective:

Secondary study objectives were to investigate the safety and efficacy of a treatment change to insulin glargine in ICT treated subjects in terms of:

* Percentage of blood glucose measurements(CGMS data)smaller/equal 60mg/dl [3.3 mmol/l].
* Percentage of nocturnal blood glucose measurements(CGMS data)smaller/equal 60mg/dl[3.3 mmol/l].
* Percentage of daytime blood glucose measurements(CGMS data)smaller/equal 60mg/dl[3.3 mmol/l].
* Area under the curve (AUC smaller/equal 60)and time(t smaller/equal 60)for blood glucose smaller/equal 60mg/dl[3.3mmol/l], area under the curve (AUC greater/equal 180)and time (t greater/equal 180) for blood glucose greater/equal 180mg/dl[10.0mmol/l].
* Area under the curve (AUC smaller/equal 60)and time(t smaller/equal 60)for blood glucose smaller/equal 60mg/dl[3.3mmol/l]during the day (AUC 06.00am - 10.00pm)and during the night(AUC 10.00pm - 06.00am).
* Area under the curve (AUC greater/equal 180)and time(t greater/equal 180)for blood glucose greater/equal 180mg/dl[10.0mmol/l]during the day (AUC 06.00am - 10.00pm)and during the night(AUC 10.00pm - 06.00am).
* Frequency of subjects with nocturnal blood glucose value smaller/equal 60mg/dl[3.3 mmol/l].
* Frequency of subjects with asymptomatic nocturnal blood glucose smaller/equal 60mg/dl[3.3 mmol/l].
* Frequency of subjects with symptomatic nocturnal blood glucose smaller/equal 60mg/dl [3.3 mmol/l].
* Frequency of subjects with daytime blood glucose smaller/equal 60mg/dl [3.3 mmol/l].
* Frequency of subjects with asymptomatic daytime blood glucose smaller/equal 60mg/dl[3.3 mmol/l].
* Frequency of subjects with symptomatic daytime blood glucose smaller/equal 60mg/dl[3.3 mmol/l].
* Frequency of subjects with hyperglycemic blood glucose(greater/equal 180mg/dl,[10.0mmol/l]).
* Frequency of subjects with symptomatic hypoglycemia(smaller/equal 60mg/dl [3.3mmol]).
* Frequency of subjects with severe hypoglycemia(smaller/equal 36mg/dl [2.0mmol/l]).
* Blood glucose values of 8-point profiles.
* Mean daytime & mean nocturnal blood glucose of 8-point-profiles.
* HbA1c.
* Fasting blood glucose (FBG).
* Dose of insulin.
* Adjustment of insulin.
* Body weight, body mass index.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with type 2 diabetes mellitus (no history of ketoacidosis)and stable treatment with NPH insulin(once or twice daily)and mealtime insulin for at least 3 months.
* HbA1c values smaller/equal 8.0%(measured at screening visit, Visit 1).
* Ability and willingness to perform continuous and self monitoring blood glucose profiles, using a self monitoring blood glucose meter as well as carrying the continuous blood glucose meter at least two times for 72 hours throughout the study at home.

Exclusion Criteria:

* All forms of diabetes other than type 2 diabetes mellitus.
* Oral antidiabetic drugs(OADs)and/or insulins other than NPH and mealtime insulins, except metformin(stable dose for a minimum of 3 months, no dose adjustments during the study).
* Pregnant(as determined by urine pregnancy test at Visit 1)or breast-feeding.
* Women of childbearing potential who did not take adequate contraceptive protection such as systemic hormones or who planned to become pregnant during the study.
* Likelihood of requiring treatment during the study period with drugs not permitted by the study protocol (e.g. systemic corticosteroids).
* History of hypersensitivity to the study medication or to drugs with similar chemical structures.
* Treatment with any investigational drugs in the last month before study entry.
* History of drug or alcohol abuse.
* Diabetic retinopathy with surgical treatment (laser photocoagulation or vitrectomy) in the 3 months prior to study entry or which required surgical treatment within the study.
* Clinically relevant cardiovascular, gastrointestinal, hepatic, neurological, endocrine, hematological or other major systemic diseases making implementation of the protocol or interpretation of the study results difficult.
* Known impaired hepatic or renal function.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480
Dates: Start 2003-10; Primary Completion 2004-03 (Actual); Study Completion 2004-03 (Actual)

PRIMARY OUTCOMES:
Frequency of subjects with conventionally detected hypoglycemia

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Landgraf, Dr., Study Director — Sanofi

REFERENCES:
- [Result] Zick R, Petersen B, Richter M, Haug C; SAFIR Study Group. Comparison of continuous blood glucose measurement with conventional documentation of hypoglycemia in patients with Type 2 diabetes on multiple daily insulin injection therapy. Diabetes Technol Ther. 2007 Dec;9(6):483-92. doi: 10.1089/dia.2007.0230. PMID 18034602